CLINICAL TRIAL: NCT05935293
Title: Impact of Continuous Perioperative Dexmedetomidine Infusion on Postoperative Renal Function Among Patients Undergoing Kidney Transplantation: a Randomized Controlled Trial
Brief Title: Dexmedetomidine and Kidney Transplantation
Acronym: DexTR
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Eduardo Schiffer (Other)
Responsible Party: Sponsor-Investigator, Eduardo Schiffer, Professor, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Dex Renal Transp
Record Dates: First submitted 2023-05-31; First posted 2023-07-07 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2023-07

CONDITIONS: Renal Transplantation; Dexmedetomidine
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine (Experimental): Patients in the dexmedetomidine group will receive intraoperative dexmedetomidine initiated in the operating room, before anesthetic induction.
  Bolus of 0.6/mcg/Kg 15 mins before induction, followed by a continuous infusion of 0.4 mcg/kg/h during the per-operative period until transfer to intensive care and then 0.1 mcg/kg/h continued for additional 24 hours.
  Interventions: Drug: Dexmedetomidine
- Control (Placebo Comparator): Patients in the control group will receive intraoperative sodium chloride 0.9% initiated in the operating room, before anesthetic induction.
  IV administration rate will be weight adapted and similar to that of Dexmedetomidine group in volume (mL) and time (minutes) Bolus of 0.6/mcg/Kg 15 mins before induction, followed by a continuous infusion of 0.4 mcg/kg/h during the per-operative period until transfer to intensive care and then 0.1 mcg/kg/h continued for additional 24 hours.
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — iv administration dexmedetomidine
  Other Names: DEX

SUMMARY:
Dexmedetomidine, an alpha 2 agonist, is being increasingly used in recent years for the maintaining of anesthesia as it allows sedation and analgesia with only a modest respiratory depression effect when compared to opioids and inhaled anesthetic agents and allows maintenance of spontaneous ventilation. Most common side effects are bradycardia and hypotension. Drug's metabolism is exclusively hepatic and therefor do not require dosage adaptation for patient's kidney function.

Post-Operative acute kidney injury (AKI) is a common complication after major surgery and might incur serious adverse outcomes such as longer hospital stay, dialysis, chronic kidney disease and death. The most common theory for the occurrence of post-operative AKI is the ischemic-reperfusion syndrome.

Several in vitro animal studies as well as human studies have suggested the nephroprotective effects of per-operative continuous infusion of dexmedetomidine and its ability to decrease post-operative AKI.

Kidney transplantation (KT) is the treatment of choice for patients with End Stage Renal Disease. It is considered a major surgery and it was shown that optimized perioperative management could improve post-operative outcomes such as early graft function as measured by urine output and serum creatinine trends. However, delayed graft function (DGF), which is defined by the need for dialysis within the first seven days after transplantation remains a significant issue for post-operative KT care with an incidence of up to 30%.

A retrospective study of 780 patients receiving KT, has shown that preoperative dexmedetomidine could significantly decrease occurrence of DGF. Recently, two single-center, randomized controlled trials, with similar sample sizes of 104 and 111 patients, compared peri-operative continuous infusion of dexmedetomidine to placebo. One study failed to show significant impact on DGF incidence while the second showed a significant 50% reduction in DGF in the dexmedetomidine group. Due to increasing evidence concerning the nephroprotective effects and improved post-operative outcomes of perioperative continuous dexmedetomidine infusion, a larger, multi-center randomized-controlled trial to study and potentially confirm the evidence in the settings of KT would be of benefit.

The aim of our study is to assess whether the perioperative continuous infusion of dexmedetomidine during KT could improve peri-operative renal function among KT recipients as compared to placebo.

DETAILED DESCRIPTION:
Study design

* Study type

  o Multi-center, Double blinded, placebo controlled, randomized trial
* Primary and secondary outcomes

  * Primary outcomes Difference in mean kinetic GFR at post operative day (POD) 1 between intervention and control group.
  * Secondary outcomes Incidence of DGF Per- and post-operative urine output Post-operative creatinine levels Time with hypotension <30% of pre-induction value Mean and median intraoperative norepinephrine Incidence of bradycardia requiring emergency treatment intraoperatively Amount of fluid administered intraoperatively Levels of renal function bio-markers (see table 1) on POD 1-2-3 Incidence of pathological radiological findings on post-operative renal ultrasound at POD 1 Evaluation of the evolution of cytological parameters of the grafts in the two groups Incidence of graft rejection during the first year after the transplantation Length of hospital and IMC/ICU stay Incidence of respiratory complications
* Population

  o After approval from the Ethics Commission of the Canton of Geneva, and after obtaining the consent of the patients, the investigators will include in the study all patients admitted for renal transplantation according to the following criteria in the study: Inclusion criteria

  a. Elective and urgent renal transplantation for end-stage renal insufficiency. Exclusion criteria
  1. Age < 18 years old
  2. Any known allergy or hypersensitivity to dexmedetomidine or clonidine
  3. Preoperative bradycardia with heart rate <50
  4. Second or third-degree atrioventricular block
  5. Left ventricular ejection fraction <30%
  6. Preoperative severe systolic dysfunction (LVEF<30%)
  7. Conduction disorders of the Mobitz 2 or Mobitz 3 type in the absence of a pacemaker
  8. Exposure to Dexmedetomidine in the past 30 days
  9. Recent cerebrovascular pathology (< 3 month)
* Data collection and measurements o Baseline data: Age, sex Months on waiting list Diabetes status Hypertension status Donor baseline creatinine and eGFR Recipient baseline creatinine and eGFR (if available)

DESCRIPTION OF STUDY PROCEDURES

Per- and Post-operative Urine Output This is a routine standard of care and will be assessed during and after the surgery daily and will allow to monitor kidney function assessing the response to the study drug Urine sample This is a routine standard of care. This will be performed before, during and after surgery to assess kidney function and reactions to given diuretics. This will allow the investigators to monitor different factors permitting better understanding of responses to the study drug.

Blood sample This is a routine standard of care and will be taken during and after the surgery (day 1 to 7 during the participants stay, then 1 and 6 months after and finally 1 year after the surgery) and will allow the investigators to monitor body's reaction to given drugs, kidney and heart function and monitor for any adverse reactions from administered drugs.

The investigators will use it to monitor different factors (including renal function bio-markers) to assess the status of the new kidney and reactions to the study drug.

Graft ultrasound This is a noninvasive procedure and the routine standard of care. Ultrasound of kidney graft will be done every post-operative day until proof of adequate graft function.

Graft biopsy This is a routine procedure and the standard of care after kidney transplantation. This will be done once during the operation, after graft reperfusion and at 6 months post transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Elective and urgent renal transplantation for end-stage renal insufficiency

Exclusion Criteria:

* Age < 18 years old
* Any known allergy or hypersensitivity to dexmedetomidine or clonidine
* Preoperative bradycardia with heart rate <50
* Second or third-degree atrioventricular block
* Left ventricular ejection fraction <30%
* Preoperative severe systolic dysfunction (LVEF<30%)
* Conduction disorders of the Mobitz 2 or Mobitz 3 type in the absence of a pacemaker
* Exposure to Dexmedetomidine in the past 30 days
* Recent cerebrovascular pathology (< 3 month)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Kinetic GFR | 30-days
  The main outcome of the study is a significant increase in GFR kinetic values on postoperative day 1 (POD1) between the intervention and control groups after continuous perioperative infusion of dexmedetomidine.

SECONDARY OUTCOMES:
Impact of dexmedetomidine on delayed graft function assessing kGFR | 1-year
  Kidney glomerular filtration rate (kGFR, mL/min)
Impact of dexmedetomidine on delayed graft function assessing GFR EPI | 1-year
  Estimated glomerular filtration rate (GFR EPI, mL/min)
Impact of dexmedetomidine on delayed graft function monitoring serum creatinine levels | 1-year
  Serum creatinine levels (ml/dL)
Impact of dexmedetomidine on delayed graft function evaluating urine output | 1-year
  Urine output (mL).
Impact of dexmedetomidine on renal glomerular biomarkers | 3-days
  Cystatin C (mg/L)
Impact of dexmedetomidine on renal structural biomarkers | 3-days
  Plasmatic NGAL (ng/mL).
Impact of dexmedetomidine on post-operative outcome. | 1-year
  Length of hospital and ICU stay (days)
Impact of dexmedetomidine on general post-operative complications. | 1-year
  Dindo-Clavien classification (grade I to V)